CLINICAL TRIAL: NCT07149168
Title: Role of Pericapsular Nerve Block Using Dexmedetomidine and Bupivacaine in Improving the Outcome of Patients Undergoing Hip Surgery Under Spinal Anesthesia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FMASU MS 760/2024
Record Dates: First submitted 2025-08-23; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2024-12

CONDITIONS: Pain During Spinal Positioning
MeSH Terms: interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): patients will recieve For spinal anesthesia in fracture neck femur surgery, a typical dose of 0.5% hyperbaric bupivacaine ranges from 0.1 to 0.15 mg/kg (2 to 3 mL), depending on the patient's height and clinical condition. Lower doses are used for shorter or elderly patients, while taller patients may require higher doses to achieve the desired block level at T10-T12
  Interventions: Drug: Bupivacain
- group B (Active Comparator): Patients in this group will first receive a pericapsular nerve block (PENG) before spinal anesthesia.
  The PENG block will be performed using a mixture of 0.25% bupivacaine (1.25 to 2.5 mg/kg.) combined with dexmedetomidine at a dose of 1.25 mcg/kg. This combination provides prolonged analgesia, enhances block effectiveness, and minimizes motor blockade, ensuring optimal pain control for fracture neck femur surgery.
  Following the successful administration of the PENG block, spinal anesthesia will be administered as described for Group A.
  Interventions: Drug: Dexmedetomidin

INTERVENTIONS:
Drug: Dexmedetomidin — The PENG block will be performed using a mixture of 0.25% bupivacaine (1.25 to 2.5 mg/kg.) combined with dexmedetomidine at a dose of 1.25 mcg/kg
  Arms: group B
Drug: Bupivacain — a typical dose of 0.5% hyperbaric bupivacaine ranges from 0.1 to 0.15 mg/kg (2 to 3 mL), depending on the patient's height and clinical condition. Lower doses are used for shorter or elderly patients, while taller patients may require higher doses
  Arms: control

SUMMARY:
the investigators will compare the effectiveness and safety of the pericapsular nerve block (PENG) using dexmedetomidine and bupivacaine before giving spinal anesthesia in improving the quality and success rate of spinal anesthesia for Fracture Neck Femur surgery versus spinal anesthesia alone.

DETAILED DESCRIPTION:
- Pre-operative settings: Patients scheduled for Fracture Neck Femur surgery under spinal anesthesia will be thoroughly evaluated pre-operatively. A detailed medical history will be obtained, and all patients will undergo a comprehensive physical examination, with particular attention to neurological assessment to exclude any pre-existing conditions that might influence the study outcomes. Additionally, pre-operative laboratory tests, including complete blood count, and coagulation profile, will be reviewed to ensure patient eligibility and safety.

2- Intraoperative Settings: Monitoring: Upon entering the operating room, standard monitoring will be applied to all patients, including pulse oximetry (SpO2), non-invasive blood pressure (NIBP), heart rate (HR), and electrocardiogram (ECG). Baseline measurements will be recorded before any anesthetic intervention.

Intravenous Access: An intravenous (IV) cannula will be inserted, and IV fluids will be initiated.

Group A (Control Group):

For spinal anesthesia in fracture neck femur surgery, a typical dose of 0.5% hyperbaric bupivacaine ranges from 0.1 to 0.15 mg/kg (2 to 3 mL), depending on the patient's height and clinical condition. Lower doses are used for shorter or elderly patients, while taller patients may require higher doses to achieve the desired block level at T10-T12.

Group B (PENG Block Group):

Patients in this group will first receive a pericapsular nerve block (PENG) before spinal anesthesia.

The PENG block will be performed using a mixture of 0.25% bupivacaine (1.25 to 2.5 mg/kg.) combined with dexmedetomidine at a dose of 1.25 mcg/kg. This combination provides prolonged analgesia, enhances block effectiveness, and minimizes motor blockade, ensuring optimal pain control for fracture neck femur surgery.

Following the successful administration of the PENG block, spinal anesthesia will be administered as described for Group A.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years, scheduled for elective fracture neck femur surgery, • Physical status: ASAI-III.

Exclusion Criteria:

* • Patients with contraindications to spinal anesthesia or regional blocks as:

  * significant coagulopathy
  * Known allergies to drugs used (Bupivacaine or dexmedetomidine)
  * Infection at site of injection

    * ASA IV
    * Cardiac patients with significant valve stenosis or sever pulmonary hypertension

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
The success rate of achieving adequate spinal anesthesia. | from injection to 24 hr post operative

CONTACTS AND LOCATIONS:
Overall Officials: Dina Sameer Ahmed AboRaya, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all data will be shared once study is completed
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: before 1/2026
Access Criteria: free